CLINICAL TRIAL: NCT00509730
Title: Multicentered Randomized Controlled Trail to Test the Cost Effectiveness of Urodynamics in Women With Symptoms of Stress Urinary Incontinence in Whom Surgical Treatment is Considered
Brief Title: Value of Urodynamics Prior to Stress Incontinence Surgery
Acronym: VUSIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: NL14625.091.06; 80-007022-98-07203
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2008-06

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; urodynamics; randomized clinical trial; surgery
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Urodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Urodynamics

SUMMARY:
To test the value of preoperatively performed urodynamics with regard to outcome of surgery for stress urinary incontinence (SUI) and to examine whether not performing urodynamics preoperatively is more cost effective than performing urodynamics preoperatively using the non-inferiority assumption.

DETAILED DESCRIPTION:
Design: multidisciplinary and multicentre randomized controlled trial

Study population/inclusion criteria : all women, not previously operated for stress incontinence, seeking help for urinary stress incontinence where conservative therapy in particular physiotherapy has failed and are opting and candidates for surgical therapy will be asked to participate in our study. Incontinence must have been demonstrated on physical examination and/or micturition diary. Patients can be included by gynaecologists or urologists who are cooperating in the study.

Intervention: consists of the non performance of urodynamics in the studygroup. The control group will undergo urodynamics as is at present the norm.

In all patients the next items will be recorded at inclusion:

1. History and clinical examination
2. 48h-Bladder(voiding and incontinence) diary,
3. 48h-Pad test
4. Validated Quality of Life questionnaires (SF 36, Euroqol 5D, UDI, IIQ)
5. Urinalysis for the detection of urinary tract infection.
6. Residual urine measured by ultrasound.

At this point an interim decision will be made for surgery. At that moment patients are informed about the study. After obtaining informed consent the patients are randomly assigned to undergo urodynamic testing or not. In the study group the decision for intervention will be based on the history and clinical examination only and will be the same as the interim decision which is surgery.

In the control group this decision will be based on history and clinical examination IN COMBINATION with the result of the urodynamic testing. It can be a decision to proceed with surgery (estimated at 2/3rd of the women) or conservative usually medication. The T0(moment of intervention) is defined as the moment of the first intervention which is by definition surgery in the study group and either surgery or conservative in the control group. After the intervention additional therapy is possible in both arms.

The follow-up period will be 24 months after T0 , in which the same parameters as pre-operative will be assessed.

These items will be assessed at:

6 weeks post intervention (PI) 3 months PI 6 months PI 12 months PI 24 months PI

Urodynamics, in the control group, will be performed according to ICS standards and consist of free flow, fillingscystometry, pressure flow study and a urethral pressure profilometry in rest and during stress. The outcomes will be matched to urodynamic findings to indicate the possible useful parts of the urodynamic findings.

Post operative urodynamics is NOT part of the study.

The primary outcome of this study is the improvement of Urogenital Distress Inventory (UDI) at 24 months after baseline and the power calculation is performed using the non-inferiority assumption. The mean improvement in UDI in both groups is expected to be 35 with standard deviation 10.(22) A difference in mean improvement of 8 or less is considered non-inferior. As this condition is allowed for one third of the total group (those women in the non-UDI group, who would not have been operatively treated), this results in a difference in mean improvement of 2.7 or less between the UDI and non-UDI group. Then effectively 130 women in each group are needed to reach a power of 70% using one-sided testing at 0.05. Considering an expected percentage lost to follow up of ca. 10%, in total 290 women (145 in each group) will be included in this study.

Multivariate analysis of covariance with group, centre and the baseline covariate as independent variables will be used to estimate differences in improvement of the UDI after 24 months between the groups with 95% confidence intervals. As the UDI is skewed, data will be logtransformed prior to analysis. Other variables (ie Incontinence Impact Questionnaire) will be analysed similar.

Economic evaluation:

For each patient, utilisation of health care services will be recorded prospectively, using Case Record Forms, including urodynamic testing, surgery for SUI, re-operations, medical treatment for detrusor instability, care for urinary incontinence, and care for urinary retention. By multiplying these volumes of care with unit cost prices, direct medical costs incurred by SUI during the follow up period will be calculated for each patient. For unit cost prices, national guidelines will be used (CVZ, 2004). For costs of care for urinary incontinence and urinary retention, data from the literature will be used, converted to 2006 prices. We incorporated the health related quality of life questionnaire euroqol 5D in our study to be able to calculate QALYs (quality-adjusted life-years), which is a measure of health outcomes. A QALY is the change in quality of life induced by the treatment multiplied by the duration of the treatment effect and it provides the number of QALYs gained. QALYs can then be related to medical costs to arrive at a final common denominator of cost/QALY. This parameter can be used to compare the cost-effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of stress urinary incontinence and/or mixed urinary incontinence, predominantly stress incontinence
* Signs of stress urinary incontinence on physical examination or voiding-diary
* Patient is a candidate for surgical treatment (as based on history and physical examination)
* Patient has attended at least 3 months of physiotherapy
* Patient accepts randomisation
* Patient is capable to fill out bladder diary's, pad tests and questionnaires
* Patient understands the Dutch written and spoken language
* ASA 1 or 2

Exclusion Criteria:

* Previous incontinence surgery
* Mixed urinary incontinence, urge component is predominant
* Prolapse >= 1cm beyond the hymen on Valsalva in supine position
* Postvoid urinary residual > 150ml
* Present urinary tract infection
* The need for additional pelvic surgery (prolapse and/or hysterectomy)
* Patient is or wants to become pregnant
* Prior pelvic radiotherapy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2007-03; Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Non inferiority among the two groups as far as the improvement in the UDI at two years after treatment is concerned.

SECONDARY OUTCOMES:
Cure of incontinence as measured by the pad test and voiding diary. Complications of surgery for stress urinary incontinence, in particular re-operations and overactive bladder symptoms. Quality of life as measured by RAND-36, Euroqol and IIQ.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Vierhout, M.D. PhD., Principal Investigator — University Medical Center St. Radboud; John Heesakkers, M.D. PhD., Principal Investigator — University Medical Center St. Radboud; Suzan Broekhuis, M.D., Principal Investigator — University Medical Center St. Radboud
Locations (1):
- UMC St.Radboud, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] van Leijsen SA, Kluivers KB, Mol BW, Broekhuis SR, Milani AL, Bongers MY, Aalders CI, Dietz V, Malmberg GG, Vierhout ME, Heesakkers JP. Can preoperative urodynamic investigation be omitted in women with stress urinary incontinence? A non-inferiority randomized controlled trial. Neurourol Urodyn. 2012 Sep;31(7):1118-23. doi: 10.1002/nau.22230. Epub 2012 Apr 6. PMID 22488817